CLINICAL TRIAL: NCT06996028
Title: Comparative Effects of (LIFT) Lower-extremity Functional Training and (PEDALS) Pediatric Endurance and Limb Strengthening on Balance and Mobility in Children With Cerebral Palsy
Brief Title: LIFT & PEDALS on Balance and Mobility in Children With CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/25/aniqa feroz
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: CP
Keywords: CP; LIFT; 6 min walk test; GMF88

STUDY DESIGN:
Intervention Model Description: A Randomized clinical trial performed,in which 20 CP children with the age of 6-12 years will be taken randomly after screening and meeting inclusion criteria. Children will be divided in two groups. Group 1 will receive LIFT for 2 hours 5 days a week. Group 2 will receive PEDALS for 2 hours 5 days a week. Pre values were taken at 1st week and then after 4th week mid values of interventions will be taken and post values of intervention will be taken after 6 weeks of intervention to measure the effects of both therapies.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The experimental group will follow the LIFT (Lifestyle Intervention for Function and Training) program, which includes exercises across four domains: strengthening (sit-to-stand, step-ups, vertical jumping, stair climbing), balance (tandem walking, one-leg standing, balancing on unstable surfaces), gait (bridging, clamshells, heel rises), and coordination (ball kicking, hopping through squares, galloping/skipping). The training will be conducted for 2 hours per day, 5 days a week, over 6 weeks . Each 2-hour session can be divided into two 1-hour sessions or four 30-minute sessions.
  Interventions: Other: Strengthening domain, Balance domain, Coordination domain, Gait domain; Other: Lower extremity strengthening, Cardiorespiratory endurance
- Group B (Experimental): Experimental Group (Group B): The PEDALS program involves stationary cycling three times a week for 30 minutes per session, divided into two phases. Phase 1 focuses on lower-limb strengthening, where participants are properly positioned on the bike and encouraged to pedal with increasing resistance as tolerated. Phase 2 targets cardiorespiratory endurance, aiming to gradually increase cycling duration to 15-30 minutes, followed by a cool-down with low-intensity pedaling until heart rate returns close to baseline.
  Interventions: Other: Strengthening domain, Balance domain, Coordination domain, Gait domain; Other: Lower extremity strengthening, Cardiorespiratory endurance

INTERVENTIONS:
Other: Strengthening domain, Balance domain, Coordination domain, Gait domain — The experimental group will engage in a structured exercise program targeting strength, balance, gait, and coordination. Strength exercises include sit-to-stand, step-ups, vertical jumping, and stair climbing. Balance training involves tandem walking, one-leg standing, and balancing on unstable surfaces. Gait exercises include bridging, clamshells, and heel rises, while coordination activities involve ball kicking, hopping through squares, and galloping/skipping. The program runs for 2 hours per day, 5 days a week, over 6 weeks, with sessions optionally split into shorter segments.
Other: Lower extremity strengthening, Cardiorespiratory endurance — Group B will follow the PEDALS program, involving stationary cycling three times a week for 30 minutes per session. Each session includes lower-limb strengthening with gradual resistance progression and cardiorespiratory endurance training aimed at increasing cycling duration to 15-30 minutes. Proper bike setup and participant support are ensured, and each session ends with a cool-down period of pedaling without resistance until heart rate returns near baseline.

SUMMARY:
Children with cerebral palsy (CP) have impaired balance due to poor postural control and coordination, increasing fall risk and limiting daily activities. This randomized controlled trial aims to compare the effects of Lower-Extremity Functional Training (LIFT) and Pediatric Endurance and Limb Strengthening (PEDALS) on balance and mobility in children with diplegic CP. A total of 22 children (ages 6-12) from Adil Special School, Sargodha, will be randomly assigned to two groups. One group will perform exercises targeting strength, coordination, gait, and balance; the other will perform pedaling exercises. Pre- and post-intervention assessments will include the 6-Minute Walk Test, GMFM-88, and Pediatric Balance Scale. Data will be analyzed using SPSS 23

DETAILED DESCRIPTION:
Balance in children with CP is impaired by poor postural control mechanism. Earlier studies on balance have found that children with CP had poor static and dynamic balance reactions than those of typically developing children . These balance problems increase risk of falls, which further affected children with cerebral palsy in performance of activities of daily living mobility and participation. Cerebral palsy also causes coordination problems. Brain can not properly send messages to muscles about how to move in smooth and well coordinated ways. The aim of the study is to analyse comparative effects of (LIFT) lower-extremity functional training and (PEDALS) pediatric endurance and limb strenghtening on balance and mobility in children with cerebral palsy The current study will be randomized control trial; data will be collected from Sargodha Adil Special School and Rehabilitation Centre.The study will include 22 patients equally divided in two groups and randomly allocated. Inclusion criteria for the study will be ability to walk independently, ability to follow 2-step instructions and complete testing. Age between 6 and 12 years. Ability to participate in group training program and children with diplegic cerebral palsy. Patients with cognitive delay,visual problems. Seizures, or if there is change in medication will be expected during the study or if patient is suffering from disease that interfered with physical activity will be excluded from the study. One experimental group will perform 4 domains of exercises (strengthening, coordination, gait and balance). In second experimental group pedalling exercise will be performed. Data collection will be done before and after intervention. Tools used for data collection will be 6 minute walk test, GMFM88, Pediatric balance scale. Data will be analysed through SPSS version 23.00.

ELIGIBILITY:
Inclusion Criteria:

* Gross Motor Function Classification System level of I to II
* Ability to follow 2-step instructions and complete testing.
* Age between 6 and 12 years.
* Children with cerebral palsy

Exclusion Criteria:

* Cognitive delay preventing 2-step instructions
* Visual problem preventing performance of interventions.
* Caregivers unable to commit to duration of intervention.
* If patient had unstable seizures.
* If any change in medication was expected during the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-29 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
6 MINUTE WALK TEST FOR ENDURANCE | Baseline, 4th week, 6th week
  The Six-Minute Walk Test (6MWT), introduced by the American Thoracic Society in 2002, is a submaximal test used to assess aerobic capacity and endurance by measuring the distance walked in six minutes.
PEDIATRIC BALANCE SCALE(BBS) | Baseline, 4th week, 6th week
  The Pediatric Balance Scale (PBS) is a modified version of the Berg Balance Scale,
  to assess balance in school-age children with mild to moderate motor impairments.
  The Pediatric Balance Scale (PBS) is a modified version of the Berg Balance Scale, designed to assess balance in school-age children with mild to moderate motor impairments. It has demonstrated strong reliability and validity, with an intraobserver ICC of 0.927, a Cronbach's alpha of 0.857, and a concurrent validity of r = 0.692 (p < 0.0005).
  The Pediatric Balance Scale (PBS) is a modified version of the Berg Balance Scale, designed to assess balance in school-age children with mild to moderate motor impairments. It has demonstrated strong reliability and validity, with an intraobserver ICC of 0.927, a Cronbach's alpha of 0.857, and a concurrent validity of r = 0.692 (p < 0.0005).

CONTACTS AND LOCATIONS:
Overall Officials: Aniqa Feroz, MS, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Asif Javed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biyik KS, Gunel MK, Akyuz EU. How does treadmill training contribute to botulinum toxin application plus routine physical therapy in ambulatory children with spastic bilateral cerebral palsy? A randomized controlled trial. Ir J Med Sci. 2023 Feb;192(1):209-217. doi: 10.1007/s11845-022-02960-9. Epub 2022 Feb 27. PMID 35224682